CLINICAL TRIAL: NCT06017102
Title: Difference in Aerosol-generating Amount Between Wired Magnetic-assisted Capsule Endoscopy System and Esophagogastroduodenoscopy Examination of Varices in Biliary Atresia Patients
Brief Title: Wired Magnetically Assisted Capsule Endoscopy and Esophageal Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Insight Medical Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202210059DIPA
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Varices
Keywords: upper endoscopy; biliary atresia
MeSH Terms: conditions — Esophageal and Gastric Varices; Biliary Atresia | interventions — Endoscopy; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wired magnetic assisted capsule endoscopy (Experimental)
  Interventions: Device: wired magnetic assisted capsule endoscopy
- esophagogastroduodenoscopy (Other)
  Interventions: Device: esophagogastroduodenoscopy

INTERVENTIONS:
Device: wired magnetic assisted capsule endoscopy — once
  Arms: wired magnetic assisted capsule endoscopy
Device: esophagogastroduodenoscopy — once
  Arms: esophagogastroduodenoscopy

SUMMARY:
The goal of this clinical trial is to compare the safeness and effectiveness of traditional esophagogastroduodenoscope (EGD) and wired magnetically assisted capsule endoscopy (MACE) in the diagnosis of esophageal varices in biliary atresia (BA) patients. The main questions it aims to answer are:

* Subjects who do wired magnetically assisted capsule endoscopy do not need to open the mouths during the process, this study also want to know whether wired magnetically assisted capsule endoscopy can reduce the generation of droplets.
* Diagnostic accuracy between traditional esophagogastroduodenoscope and wired magnetically assisted capsule endoscopy in biliary atresia patients with esophageal varices.

Participants will do either traditional esophagogastroduodenoscope or wired magnetically assisted capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Biliary atresia patients > 6 years old
* Vital signs are stable
* Without acute gastrointestinal bleeding

Exclusion Criteria:

* Patients with metal implants, metal stent, artificial joints, bone plates, and bone screw
* Patients with electronic devices, such as pacemakers, cochlear implants, or other implanted electronic medical devices
* Throat or esophageal obstruction leading to dysphagia patients
* Consciousness disturbance patients unable to swallow
* Patients with acute upper gastrointestinal bleeding
* Patients with platelet lower than 40K or PT INR > 1.5

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period is from August 2023 to February 2025, conducted at the Gastroenterology Clinic of National Taiwan University Children's Hospital.
Groups:
- Wired Magnetic Assisted Capsule Endoscopy: This prospective open-label trial enrolls 25 patients aged 6 or older with biliary atresia to undergo wired magnetic-assisted capsule endoscopy (MCE) for esophageal varices, based on the patient's or family's choice.
- Esophagogastroduodenoscopy: Additionally, 25 patients aged 6 years or older with biliary atresia will undergo esophagogastroduodenoscopy for esophageal varices assessment as the control group.
Period: Overall Study
Arm/Group | Wired Magnetic Assisted Capsule Endoscopy | Esophagogastroduodenoscopy
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 50 participants completed the trial.
Groups:
- Wired Magnetic Assisted Capsule Endoscopy: Participants in this group undergo wired magnetic-assisted capsule endoscopy to assess esophageal varices, which is a non-invasive method decided based on the patient's or family's choice.
- Esophagogastroduodenoscopy: Participants in this group undergo esophagogastroduodenoscopy to assess esophageal varices, which is a traditional invasive method, with sedation based on the need.
- Total: Total of all reporting groups
Arm/Group | Wired Magnetic Assisted Capsule Endoscopy | Esophagogastroduodenoscopy | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 17.75 [13.60 to 27.10] | 11.10 [8.38 to 17.95] | 15.04 [10.65 to 23.44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 13 | 12 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body height [Median (Inter-Quartile Range); unit: cm] | 158 [151 to 170.5] | 143 [129.5 to 162] | 155 [141.5 to 165]
Body weight [Median (Inter-Quartile Range); unit: kg] | 53 [43 to 66.25] | 34.5 [28.25 to 52.15] | 50.15 [34.375 to 55.5]
Liver cirrhosis [Count of Participants; unit: Participants] | 13 | 17 | 30
Ascites [Count of Participants; unit: Participants] | 4 | 2 | 6
Splenomegaly [Count of Participants; unit: Participants] | 14 | 19 | 33
Liver transplantation [Count of Participants; unit: Participants] | 10 | 8 | 18
Conscious sedation [Count of Participants; unit: Participants] | 0 | 20 | 20
< 19 years of age [Count of Participants; unit: Participants] | 13 | 19 | 32
ALT [Median (Inter-Quartile Range); unit: IU/mL] | 22 [12.5 to 46] | 36 [14 to 81.5] | 30 [15.5 to 52.5]
Platelet [Median (Inter-Quartile Range); unit: K/uL] | 175 [107.5 to 220.5] | 104 [61.5 to 234.5] | 157.5 [75 to 228.25]
Hb [Median (Inter-Quartile Range); unit: g/dL] | 13.1 [11.1 to 15.1] | 11.9 [10.0 to 12.8] | 12.45 [11.225 to 14.225]
WBC [Median (Inter-Quartile Range); unit: K/uL] | 5.14 [3.74 to 6.54] | 4.2 [2.69 to 6.65] | 4.685 [3.43 to 6.46]
Total bilirubin [Median (Inter-Quartile Range); unit: mg/dL] | 1.14 [0.73 to 1.95] | 0.87 [0.55 to 2.15] | 0.985 [0.63 to 2.0075]
Direct bilirubin [Median (Inter-Quartile Range); unit: mg/dL] | 0.27 [0.18 to 0.76] | 0.21 [0.14 to 0.93] | 0.23 [0.17 to 0.89]

OUTCOME MEASURES:

1. Primary Outcome: Aerosol-generating Amount
Description: Aerosol-generating amount were measured using the MET ONE airborne particle counter [DR-528 Handheld Particle Counter (Met One Instruments, Inc., Grants Pass, OR)].
  The device was placed on a platform at the same horizontal level as the patient lying flat, to capture airborne particles (sizes: 0.3-10 μm).Background environmental values were measured prior to each procedure and subtracted to determine net aerosol generation. Results are expressed as the total number of particles generated.
Time Frame: 1 day
Population: All 50 participants completed the trial.
Measure: Median (Inter-Quartile Range); unit: Particles generated
Groups:
- Esophagogastroduodenoscopy: 25 patients aged 6 years or older with biliary atresia undergoing conventional esophagogastroduodenoscopy (EGD) for esophageal varices survey will be enrolled as the "control group."Both groups will prospectively enter the study after providing informed consent and signing the consent form. All patients will fast appropriately according to endoscopic examination guidelines before the procedure.Patients undergoing conventional EGD may choose to receive conscious sedation based on clinical needs.
- Wired Magnetic Assisted Capsule Endoscopy: In this study, 25 patients aged 6 years or older with biliary atresia undergoing Magnetic-Assisted Capsule Endoscopy (MACE) for esophageal varices survey will be enrolled as the "study group.Patients undergoing MACE will be advised to keep their lips closed and wear a surgical mask during the examination.
Arm/Group | Esophagogastroduodenoscopy | Wired Magnetic Assisted Capsule Endoscopy
Number analyzed (Participants) | 25 | 25
Particles generated
  0.3 μm | 8195 [0 to 95738] | 0 [0 to 57030]
  0.5 μm | 13296 [3570 to 57254] | 1483 [0 to 13233]
  1.0 μm | 11792 [3148 to 25064] | 3506 [949 to 8100]
  2.5 μm | 7042 [2784 to 14070] | 1978 [803 to 7421]
  4.0 μm | 1066 [360 to 2314] | 362 [109 to 1316]
  5.0 μm | 433 [113 to 1454] | 185 [41 to 639]
  7.0 μm | 143 [63 to 5701] | 41 [0 to 217]
  10.0 μm | 68 [0 to 632] | 0 [0 to 129]

2. Secondary Outcome: Particles Generated Per Minute
Description: The total number of particles of each size divided by examination time to calculate per-minute production; comparison between the two groups.
Time Frame: 1 day
Population: All 50 participants completed the trial.
Measure: Median (Inter-Quartile Range); unit: Particles generated per minute
Arm/Group | Esophagogastroduodenoscopy | Wired Magnetic Assisted Capsule Endoscopy
Number analyzed (Participants) | 25 | 25
Particles generated per minute
  0.3 μm per min | 1394 [0 to 13768] | 0 [0 to 4060]
  0.5 μm per min | 2060 [417 to 4713] | 1493 [0 to 1753]
  1.0 μm per min | 1366 [367 to 3466] | 221 [113 to 829]
  2.5 μm per min | 760 [230 to 2294] | 127 [60 to 548]
  4.0 μm per min | 117 [28 to 326] | 20 [7 to 83]
  5.0 μm per min | 69 [16 to 178] | 10 [2 to 38]
  7.0 μm per min | 22 [6 to 72] | 3 [0 to 16]
  10.0 μm per min | 10 [0 to 69] | 0 [0 to 14]

3. Secondary Outcome: Number of Participants With Esophageal Varices
Description: We recorded the number of participants who had esophageal varices after completion of the examination.
Time Frame: 1 day
Population: All 50 participants completed the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Esophagogastroduodenoscopy | Wired Magnetic Assisted Capsule Endoscopy
Number analyzed (Participants) | 25 | 25
Participants | 22 | 10

4. Secondary Outcome: Number of Participants With Gastric Varices
Description: We recorded the number of participants who had gastric varices after completion of the examination.
Time Frame: 1 day
Population: All 50 participants completed the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Esophagogastroduodenoscopy | Wired Magnetic Assisted Capsule Endoscopy
Number analyzed (Participants) | 25 | 25
Participants | 2 | 3

5. Secondary Outcome: Questionnaire Assessments
Description: After the procedure, we assessed the patient's pain level using a Visual Analogue Scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 indicates severe pain. We also evaluated the patient's willingness to undergo the same procedure again using a questionnaire scored from 0 to 5, where 0 indicates no willingness and 5 indicates strong willingness to repeat the procedure.
Time Frame: 1 day
Population: All 50 participants completed the trial.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Esophagogastroduodenoscopy | Wired Magnetic Assisted Capsule Endoscopy
Number analyzed (Participants) | 25 | 25
score on a scale
  Pain level | 0 [0 to 3] | 3 [1 to 4]
  Patient's willingness to undergo the same procedure again | 4 [3 to 5] | 4 [3 to 4.5]

6. Secondary Outcome: Examination Time
Description: Examination time is defined as the procedure duration, measured from insertion of the examination device into the participant's mouth to complete removal of the device.
Time Frame: 1 day
Population: All 50 participants completed the trial.
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Esophagogastroduodenoscopy | Wired Magnetic Assisted Capsule Endoscopy
Number analyzed (Participants) | 25 | 25
min | 7 [5 to 10] | 15 [9.5 to 19]

7. Secondary Outcome: Completion Rate
Description: Completion rate was defined as the proportion of participants in whom successful examination of each anatomical segment (esophagus, stomach, and duodenum) was achieved.Successful completion for each segment was defined as the device reaching and examining the target segment.
Time Frame: 1 day
Population: All 50 participants completed the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Esophagogastroduodenoscopy | Wired Magnetic Assisted Capsule Endoscopy
Number analyzed (Participants) | 25 | 25
Participants
  Esophagus | 25 | 25
  Stomach | 25 | 25
  Duodenum | 25 | 23

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on the day of the examination, up to 1 day.
Groups:
- Wired Magnetic Assisted Capsule Endoscopy: MACE will be advised to keep their lips closed and wear a surgical mask during the examination.
- Esophagogastroduodenoscopy: Patients undergoing conventional EGD may choose to receive conscious sedation based on clinical needs.
Arm/Group | Wired Magnetic Assisted Capsule Endoscopy | Esophagogastroduodenoscopy
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wired Magnetic Assisted Capsule Endoscopy (N=25) | Esophagogastroduodenoscopy (N=25)
Decreased Oxygen Saturation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — The participant experienced saliva aspiration coughing during esophagogastroduodenoscopy under anesthesia.

LIMITATIONS AND CAVEATS:
The limitation of this study is that the sample size for each group is not large. This limitation is due to the rarity of biliary atresia, with an incidence of only 1.5 cases per 10,000 in Taiwan. Additionally, since the examination equipment differs between the two groups, a double-blind design could not be implemented.Because biliary atresia cases are prone to infection and bleeding, it is not ethically appropriate to have each patient undergo both groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT06017102/Prot_SAP_000.pdf